CLINICAL TRIAL: NCT02555930
Title: Clinical Phenotyping and Genotyping of HIV-Associated Sensory Neuropathy: The HIV-POGO Study
Acronym: HIV-POGO
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 14/LO/1574
Record Dates: First submitted 2015-07-14; First posted 2015-09-22 (Estimated); Results first posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: HIV; Sensory Neuropathy; Neuropathic Pain
Keywords: HIV; Sensory Neuropathy
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No Intervention — No intervention - observational only

SUMMARY:
This study aims to recruit a cohort of HIV patients with and without HIV-SN and to identify genetic risk factors for the development of HIV-SN and neuropathic pain. It also aims to more deeply phenotype the condition, using well validated questionnaires, and to identify any influence that early neurocognitive dysfunction may have on the reporting, diagnosis and treatment of neuropathic pain in the HIV population.

DETAILED DESCRIPTION:
HIV associated sensory neuropathy (HIV-SN) is a frequent complication of HIV infection, affecting between 20 and 57% of infected individuals. The advent of better antiretroviral treatment for HIV has meant that mortality from HIV has decreased dramatically in the UK. This means however, that chronic, age-related conditions associated with HIV, such as HIV-SN and cognitive impairment, are increasing in prevalence and becoming a significant disease burden.

The classification, diagnosis and treatment of HIV-SN remains poor. Currently, little is known about the genetic basis of the disorder and what risk factors mean that some patients with HIV develop neuropathy and pain, whilst others do not. It is hoped that by further characterising or 'phenotyping' the disorder, it will be easier to identify which patients are at risk of developing neuropathy and chronic pain. It may also mean that treatment can be more individualised as currently patients often undergo a frustrating 'trial and error' protocol of treatment, as clinicians can not yet predict who will respond to which treatment.

It has also been suggested that there is a link between HIV-SN and HIV associated neurocognitive disorder (HAND), which is another common, age-related complication of HIV infection. It may be that the existence of one pathology could predict the development of the other, or that the presence of HAND may impair the diagnosis or treatment of chronic pain associated with HIV-SN.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over
* HIV infection

Exclusion Criteria:

* co-incident severe neurological disease
* co-incident severe psychiatric illness
* limited english language skills so as not able to conduct quantitative sensory testing
* pregnancy
* pain of greater than 3/10 on an NRS due to pathology other than HIV-SN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals over the age of 18 of any gender with HIV
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew SC Rice, Prof, Principal Investigator — Imperial College London
Locations (1):
- Pain Research Group, Dept Surgery & Cancer, Imperial College, Chelsea and Westminster Campus, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sipila R, Kemp H, Harno H, Rice ASC, Kalso E. Health-related quality of life and pain interference in two patient cohorts with neuropathic pain: breast cancer survivors and HIV patients. Scand J Pain. 2021 Mar 17;21(3):512-521. doi: 10.1515/sjpain-2020-0177. Print 2021 Jul 27. PMID 33725747

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: NA all recruited were included
Groups:
- Total Cohort: Observational study whole cohort - Adults with HIV infection (with or without sensory neuropathy and/or neuropathic pain)
Period: Overall Study
Arm/Group | Total Cohort
Started | 148
Completed | 148
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants recruited are included
Groups:
- Total Cohort: Observational study whole cohort - Adults with HIV infection (with or without sensory neuropathy or neuropathic pain)
Arm/Group | Total Cohort
Number analyzed (Participants) | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 123
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 117
  Black | 22
  Other | 9
Employment [Count of Participants; unit: Participants]
  Employed | 79
  Not working through illness | 41
  Unemployed | 10
  Retired | 18

OUTCOME MEASURES:

1. Primary Outcome: Neuropathic Element of Pain Using the Doleur Neuropathique 4 Interview
Description: Doleur Neuropathique 4 Interview score greater than or equal to 4, indicating a high likelihood of neuropathic pain
Time Frame: Day 1
Population: Adults with HIV infection
Measure: Count of Participants; unit: Participants
Groups:
- Total Cohort: Whole cohort - Adults with HIV infection
Arm/Group | Total Cohort
Number analyzed (Participants) | 148
Participants
  DN4 >3 | 81
  DN4 <4 | 67

2. Secondary Outcome: Cognitive Function: Global T-score for Cogstate Computerised Cognitive Function Test Set
Description: Cogstate computerised cognitive function testing. A global T-score is a composite measure determined by the arithmetric mean of 8 test scores covering the following cognitive domains: psychomotor function, visual learning, working memory, executive function, emotional recognition, verbal learning, attention and verbal memory. Raw scores were converted to a standardised T score using age adjusted normative data (mean 50; standard deviation 10). Higher scores are interpreted as 'better' cognitive function.
Time Frame: Day 1
Population: All participants that completed Cogstate cognitive function testing
Measure: Mean (Standard Deviation); unit: T-score for global measure of function
Arm/Group | Total Cohort
Number analyzed (Participants) | 140
T-score for global measure of function | 48.09 (8.07)

3. Secondary Outcome: Conditioned Pain Modulation Efficiency
Description: Conditioned Pain Modulation (CPM) efficiency to protocol using a cold noxious stimulus. The CPM efficiency is calculated as the pressure pain threshold (measured with an algometer on the forearm) during the noxious conditioning stimulus minus the pressure pain threshold prior to conditioning stimulus.
Time Frame: Day 1
Population: All subjects who completed full Conditioned Pain Modulation protocol
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Total Cohort
Number analyzed (Participants) | 63
kPa | 0.78 (0.80)

ADVERSE EVENTS:
Time Frame: Adverse data was recorded for the 24 hours following the single clinical appointment for this observational study - the study did not involve an intervention and the only invasive procedure was a venous blood sample
Groups:
- Total Cohort: Observational study whole cohort
Arm/Group | Total Cohort
All-Cause Mortality (participants affected / at risk) | 0/148
Serious Adverse Events (participants affected / at risk) | 0/148
Other Adverse Events (participants affected / at risk) | 0/148

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/30/NCT02555930/Prot_SAP_000.pdf